CLINICAL TRIAL: NCT02378896
Title: Personalized Computerized Inhibitory Control Training for OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #7059
Record Dates: First submitted 2015-02-27; First posted 2015-03-04 (Estimated); Last update posted 2018-01-29 (Actual); Status verified 2018-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Cognitive Behavioral Therapy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CBT + Personalized Computer Program (Experimental): Cognitive Behavioral Therapy (CBT), consisting of Exposure and Ritual Prevention Therapy and training with a personalized computerized inhibitory training program
  Interventions: Behavioral: Personalized Computer Program; Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Personalized Computer Program — Training with a personalized computerized inhibitory training program
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy (CBT), consisting of Exposure and Ritual Prevention Therapy

SUMMARY:
This study will evaluate the effects of a computerized training program coupled with cognitive behavioral therapy (CBT) for OCD.

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of a computerized training program (called Personalized Computerized Inhibitory Training, or PCIT) coupled with cognitive behavioral therapies (CBT) consisting of Exposures and Response Prevention in treating obsessive compulsive disorder (OCD) in patients who previously underwent CBT, but still have residual symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Principal diagnosis of OCD (assessed by SCID).
* Clinically significant OCD symptoms (Y-BOCS score of at least 16).
* Have a history of completing a trial of at least 1 EX/RP sessions.
* Have access to a computer or laptop.

Exclusion Criteria:

* Individuals with the following disorders will excluded: bipolar, psychosis, current major depressive disorder (assessed by SCID).
* Patients with head injury and loss of consciousness of more than five minutes or a neurological condition affecting the central nervous system.
* Patients taking a psychiatric medication will be asked to maintain a stable dose for 6 weeks prior to study entry.
* Vision or hearing loss (although individuals with vision corrected by glasses or contacts will not be excluded).
* Active suicidality warranting immediate clinical care.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Obsessive-compulsive symptoms measured after 3 weeks of treatment | 3 weeks
  measured by Yale Brown Obsessive Compulsive Scale (YBOCS)

CONTACTS AND LOCATIONS:
Overall Officials: Helen B Simpson, M.D., PhD, Principal Investigator — New York State Psychiactic Institute, Anxiety Disorders Clinic
Locations (1):
- New York State Psychiactic Institute, New York, New York, United States